CLINICAL TRIAL: NCT05695248
Title: A Phase 1b/2 Single and Multiple Dose Study to Assess the Safety, Tolerability, Clinical Activity, Pharmacokinetics, Pharmacodynamics, and Immunogenicity of STAR-0215 in Participants With Hereditary Angioedema (The ALPHA-STAR Trial)
Brief Title: A Study of STAR-0215 in Participants With Hereditary Angioedema
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Astria Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: STAR-0215-201; 2022-502953-32 (EudraCT Number)
Record Dates: First submitted 2023-01-06; First posted 2023-01-23 (Actual); Last update posted 2025-04-11 (Actual); Status verified 2024-07

CONDITIONS: Hereditary Angioedema
Keywords: HAE; Angioedema
MeSH Terms: conditions — Angioedemas, Hereditary; Angioedema

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (3):
- Cohort 1 - Single Dose (Experimental): Participants will receive 1 dose of STAR-0215.
  Interventions: Drug: STAR-0215
- Cohort 2 - Multiple Dose (Experimental): Participants will receive 2 doses of STAR-0215 administered 3 months apart.
  Interventions: Drug: STAR-0215
- Cohort 3 - Multiple Dose (Experimental): Participants will receive 2 doses of STAR-0215 administered 1 month apart.
  Interventions: Drug: STAR-0215

INTERVENTIONS:
Drug: STAR-0215 — STAR-0215 will be administered as a subcutaneous bolus injection.

SUMMARY:
The goal of this clinical trial is to test the drug STAR-0215 in participants with hereditary angioedema (HAE). One group of participants will get 1 dose of STAR-0215, and two other groups will get 2 doses of STAR-0215. Researchers will study the effects of STAR-0215 in participants with HAE as this is the first time that the drug has been given to participants with HAE.

DETAILED DESCRIPTION:
This is a Phase 1b/2 single and multiple dose trial evaluating the safety, tolerability, clinical activity, pharmacokinetics, pharmacodynamics, and immunogenicity of subcutaneous administration of STAR-0215 in participants with type I or type II HAE in 3 dose cohorts. The first cohort will receive 1 dose of STAR-0215; the second and third cohorts will receive 2 sequential doses. This is the first trial of STAR-0215 in participants with HAE and the first evaluation of a multiple-dose regimen. After the required follow up period, participants who are willing and eligible to consent can begin participation in the long-term open label extension study (STAR-0215-202, ALPHA-SOLAR).

ELIGIBILITY:
Inclusion Criteria:

1. Documented diagnosis of HAE (type I or II). The following must be met:

   a. Documented clinical history consistent with HAE (for example, subcutaneous or mucosal, nonpruritic swelling episodes without accompanying urticaria).
2. Experienced at least 2 HAE attacks during the Run-In period, as confirmed by an investigator based on meeting the protocol-specified definition of an HAE attack.

Exclusion Criteria:

1. Any concomitant diagnosis of another form of chronic angioedema, such as acquired C1 inhibitor deficiency, HAE with normal C1-INH (also known as HAE type III), idiopathic angioedema, or angioedema associated with urticaria.
2. Use of therapies prescribed for the prevention of HAE attacks prior to Screening:

   1. lanadelumab within 90 days
   2. berotralstat within 21 days
   3. all other prophylactic therapies, within 7 days
3. Any exposure to angiotensin-converting enzyme inhibitors or any estrogen containing medications with systemic absorption (such as hormonal contraceptives or hormone replacement therapy) within 28 days prior to Screening.
4. Any exposure to androgens (for example, stanozolol, danazol, oxandrolone, methyltestosterone, testosterone) within 7 days prior to Screening.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2023-02-21 (Actual); Primary Completion 2025-03-13 (Actual); Study Completion 2025-03-13 (Actual)

PRIMARY OUTCOMES:
Number of Participants Experiencing Treatment-emergent Adverse Events | Day 1 through Day 448 (Cohort 1), Day 531 (Cohort 2), and Day 475 (Cohort 3)

SECONDARY OUTCOMES:
Change From Baseline in Monthly HAE Attack Rate | Baseline through Day 168 (Cohort 1), Day 251 (Cohort 2), and Day 195 (Cohort 3)
Severity of HAE Attacks Experienced by Participants | Cohort 1: Day 1 through Day 168; Cohort 2: Day 1 through Day 251; Cohort 3: Day 1 through Day 195
  All HAE attacks will be classified according to severity (mild, moderate, and severe).
Duration of HAE Attacks | Cohort 1: Day 1 through Day 168; Cohort 2: Day 1 through Day 251; Cohort 3: Day 1 through Day 195
  Duration will be reported as shorter than 12 hours, 12 to 24 hours, 24 to 48 hours, and longer than 48 hours.
Number of Participants Experiencing HAE Attacks Requiring On-demand Therapy | Cohort 1: Day 1 through Day 168; Cohort 2: Day 1 through Day 251; Cohort 3: Day 1 through Day 195
Time to First HAE Attack After First and Last Dosing | Cohort 1: Day 1 through Day 168; Cohort 2: Day 1 through Day 251; Cohort 3: Day 1 through Day 195
Serum Concentration of STAR-0215 | Cohort 1: Day 1 (pre-dose, 4 hours post dose) up to Day 168; Cohort 2: Days 1 and 84 (pre-dose, 4 hours post dose) up to Day 251; Cohort 3: Days 1 and 28 (pre-dose, 4 hours post dose) up to Day 195
  Blood samples will be collected to measure the serum concentration of STAR-0215 before and after study drug administration.
Plasma Levels of Cleaved High-molecular-weight Kininogen | Cohort 1: Day 1 (pre-dose, 4 hours post dose) up to Day 168; Cohort 2: Days 1 and 84 (pre-dose, 4 hours post dose) up to Day 251; Cohort 3: Days 1 and 28 (pre-dose, 4 hours post dose) up to Day 195
  Blood samples will be collected to measure the plasma levels of cleaved high-molecular-weight kininogen (a measure of plasma kallikrein activity).
Number of Participants with Anti-drug Antibodies To STAR-0215 | Cohort 1: Day 1 (pre-dose); Days 14, 28, 56, 84, 112, 140, and 168; Cohort 2: Days 1 and 84 (pre-dose); Days 14, 28, 56, 111, 167, and 251; Cohort 3: Days 1 and 28 (pre-dose); Days 14, 55, 111, and 195
  Blood samples will be collected to assess the formation of STAR-0215 anti-drug antibodies in serum before and after study drug administration.

CONTACTS AND LOCATIONS:
Locations (20):
- United States (13):
  - Allervie Clinical Research, Birmingham, Alabama
  - Medical Research of Arizona a Division of Allergy, Asthma & Immunology Associates, LTD., Scottsdale, Arizona
  - Allergy & Asthma Clinic of Northwest Arkansas, Bentonville, Arkansas
  - Acuro Research, Inc., Little Rock, Arkansas
  - UC San Diego US HAEA Angioedema Center, San Diego, California
  - Raffi Tachdjian MD, Inc, Santa Monica, California
  - Allergy & Asthma Clinical Research, Walnut Creek, California
  - Institute for Asthma and Allergy, PC, Chevy Chase, Maryland
  - Massachusetts General Hospital, Boston, Massachusetts
  - Washington University School of Medicine, St Louis, Missouri
  - Optimed Research, Columbus, Ohio
  - Penn State Health Milton S. Hershey Medical Center, Hershey, Pennsylvania
  - AARA Research Center, Dallas, Texas
- Diagnostical Consultative Center Convex Ltd., Sofia, Bulgaria
- Canada (2):
  - University of Alberta, Edmonton, Alberta
  - Ottawa Allergy Research Corporation, Ottawa, Ontario
- Institute of Clinical Immunology/Allergology, Faculty Hospital, Hradec Králové, Czechia
- Charité Universitätsmedizin Berlin, Berlin, Germany
- United Kingdom (2):
  - Addenbrooke's Hospital, Cambridge
  - St. James's Hospital, Leeds

IPD SHARING:
Plan to Share IPD: No